CLINICAL TRIAL: NCT04950855
Title: Evaluation of Retinal and Choroidal Microvascular Structures: Comparison With Three Trimesters of Healthy Pregnant Women and Healthy Non-pregnant Women Using Optical Coherence Tomography Angiography
Brief Title: Retinal and Choroidal Microvascular Changes During Pregnancy Period Detected With Optical Coherence Tomography Angiography
Status: Terminated | Type: Observational
Why Stopped: Due to the difficulty in following pregnant women due to the covid 19 pandemic
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Çisil Erkan Pota, Medical Doctor, Akdeniz University
Other Study IDs: Study1
Record Dates: First submitted 2021-06-24; First posted 2021-07-06 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Tomography, Optical Coherence; Choroid; retina
MeSH Terms: interventions — Tomography, Optical Coherence; Corneal Pachymetry; Tonometry, Ocular; Blood Pressure Determination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: Healty pregnant women between 18-45 years,with no history of eye surgery and systemical disease.In 1st , 2nd and 3rd trimesters the measurements will be repeated
  Interventions: Diagnostic Test: Optical Coherence Tomography,Optical Coherence Tomography Angiography(Topcon)
- Control Group: Healty non-pregnant women between 18-45 years with no history of eye surgery and systemical disease.
  Interventions: Diagnostic Test: Optical Coherence Tomography,Optical Coherence Tomography Angiography(Topcon)

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography,Optical Coherence Tomography Angiography(Topcon) — Optical coherence tomography optical coherence tomography angiography
  Other Names: Pachymetry; Otorefractometry; Tonometry; Blood Pressure Measurement

SUMMARY:
During pregnancy many physiological changes and adaptations occur.Hormonal, hematological and hemodynamic changes are responsible for most of the ocular adaptations.We are planning to compare the choroid and retinal blood flow values and choroidal thickness of pregnant women and healthy non pregnant women with optical coherence tomography and optic coherence tomography angiography

DETAILED DESCRIPTION:
During pregnancy many physiological changes and adaptations occur such as pulmonary, renal, endocrinological, haematological and visual system changes are happening. In previous studies, retinal and choroidal pregnancy-related changes in blood flow and choroidal thickness have been demonstrated. Optical coherence tomography angiography (OCTA) detects the contrast of motion in the blood flow, detecting the capillary of the retina and choroid.

It is a new functional method that visualizes the retinal networks and outer retina without using dyes.It is a non-invasive method that provides volumetric angiography information. In this study evaluation of the variability of choroidal and retinal blood flow changes and choroidal thickness, between trimesters of pregnancy and the non-pregnant control group is planned. Choroid and Retinal Blood Flow Values and Choroidal thickness in 41 pregnant women in the first trimester and it would be repeated at second and third trimesters. We compare measured values between trimesters and 45 healthy non-pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women Age > 18 years

Exclusion Criteria:

* Systemical disease such as diabetes mellitus or hypertension
* Refractive error; spherical equivalence > 4 diopters
* Ocular disease or surgery history

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Retinal and choroid thickness and retinal angiographic values will be measured in healthy pregnant population (1 time for each trimester,totally 3 times) and healty control group
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | 40 weeks
  Choroidal thickness is measured by optical coherence tomography
Retinal thickness | 40 weeks
  Retinal thickness is measured by optical coherence tomography

SECONDARY OUTCOMES:
Foveal avascular zone(FAZ) area measurement | 40 weeks
  FAZ area is measured by optical coherence tomography anjiography
Retinal vascular density | 40 weeks
  % of retinal vascular density is measured by optical coherence tomography angiography
Retinal nerve fiber layer thickness | 40 weeks
  Retinal nerve fiber layer thickness (um) is measured by optical coherence tomography
Ganglion cell layer measurement | 40 weeks
  Ganglion cell layer measurement is measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes